CLINICAL TRIAL: NCT02257905
Title: A Non-interventional Prospective Study on Allogeneic Stem Cell Transplantation in Patients With AL Amyloidosis
Brief Title: Allo SCT in Amyloidosis Non-interventional Study
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: 42206633
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: AL Amyloidosis
Keywords: AL Amyloidosis; Amyloidosis; allogeneic; HSCT
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AL Amyloidosis patients who received allo HSCT

SUMMARY:
Light-chain (AL-) amyloidosis is a very rare monoclonal plasma cell disorder with poor prognosis. Rarity of disease has precluded performance of randomized controlled trials comparing various possible treatment modalities. In general, treatment of AL amyloidosis has been adapted from myeloma (MM) therapy. There is large experience with allo SCT in MM. Based on small series of patients and case reports allogeneic transplant has emerged as potentially effective. However, more formal proof of concept of using allogeneic hematopoietic transplantation for treatment of AL Amyloidosis is lacking.

Therefore, given the limitations of conventionally collected registry data (dubious follow-up information and extreme heterogeneity), we developed the: "EBMT non-interventional prospective study on allogeneic transplantation in AL Amyloidosis" which means that transplant centers that already do perform allogeneic transplants for AL Amyloidosis will be encouraged to register their patients with AL Amyloidosis very timely with the EBMT, followed by mandatory submission of EBMT MedB and follow-up forms. The diagnosis of AL Amyloidosis would be based on uniform criteria. All EBMT centres performing allogeneic transplants for Amyloidosis will be invited to participate in this study and centres will be asked to report all AL Amyloidosis cases referred for transplantation using a simple registration form and then to submit Amyloidosis MED B forms for each transplanted patient and follow-up forms as necessary. In conclusion, it should be possible to largely improve the usual quality of registry-based data and to generate scientifically sound knowledge on HSCT in an orphan disease such as AL Amyloidosis.

DETAILED DESCRIPTION:
Short description of the study:

We plan to select those centres within the EBMT that in the past have performed any allogeneic transplant for amyloidosis and ask them to participate by completing a centre registration form. When they have a patient they want to include in this study, the centre will notify the CLWP data office of the planned allogeneic transplant the day before the transplant takes place. For this, the centre can use a patient registration form. Once a patient is included, MED B and regular follow-up are mandatory. Data entry of MED B forms and follow up will be performed in the way that is usual for the centre (either by the centre itself, by the national registry or by the Paris data office). The CLWP data office will keep track of the data submitted.

Research design:

This study is designed as a non-interventional prospective study.

Study Population:

Male or female subjects, 18 years to 60 years, with AL amyloidosis who will receive allogeneic transplantation.

Data to be collected/analysed:

The primary endpoint of this study is efficacy (best hematological remission and organ response) of allogeneic SCT in patients with AL amyloidosis. The secondary endpoints are acute and chronic GvHD, TRM and event-free and overall survival.

Purpose of the non-interventional prospective study request:

The main purpose of this non-interventional prospective study is the evaluation of the effectiveness of allogeneic transplant for AL Amyloidosis. It is planned that results will be presented on scientific symposia and that they will suffice for at least one publication (original article).

ELIGIBILITY:
Inclusion Criteria:

* AL Amyloidosis, allogeneic HSCT after November 2009, between 18-60 years at time of transplant.

Exclusion Criteria:

* other diagnoses than AL Amyloidosis, auto transplant, transplant before November 2009, younger than 18 or older than 60 at time of transplant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male or female subjects, 18 years to 60 years, with AL amyloidosis who will receive allogeneic transplantation
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-12; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
efficacy of allo sct in patients with AL Amyloidosis | 5 years
  • To evaluate the efficacy of allogeneic SCT in patients with AL Amyloidosis (best hematological remission and organ response).

SECONDARY OUTCOMES:
EFS | 5 years
  • To evaluate event-free survival.
OS | 5 years
  to evaluate overall survival

OTHER OUTCOMES:
safety of allo sct in patients with AL Amyloidosis | 5 years
  • To evaluate safety of allogeneic SCT in patients with AL Amyloidosis (TRM, incidence of acute and chronic GvHD, non-haematological toxicity and engraftment).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schoenland, MD, Principal Investigator — Medizinische Klinik, University of Heidelberg, Germany; Nicolaus Kroeger, MD, Study Chair — BMT Centre, University Hospital Eppendorf, Hamburg, Germany
Locations (4):
- CHRU Limoges, Limoges, France
- Germany (2):
  - University Hospital Eppendorf, Hamburg
  - University of Heidelberg, Heidelberg
- University Hospital, Basel, Switzerland

REFERENCES:
- [Background] Schönland et al. EBMT retrospective data, Blood 2005.
- [Background] Schönland et al. DLI data, Haematologica, 2008.